CLINICAL TRIAL: NCT05939154
Title: Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine
Brief Title: Early Identification of Mental Disorders: Application of a Multi-modal & Domains System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: CRC2021DX01
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2022-11

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mental disorders: Patients in Shanghai Mental Health Center; meet ICD-11 or DSM-5 diagnosis of depressive disorders, bipolar disorders, schizophrenia, obsessive-compulsive disorder, anxiety disorders, addictive disorders and sleep-wake disorders (do not limit subtypes and current disease state); age ≥15 years and < 60 years.
- healthy controls: Age ≥15 years and < 60 years; gender match with patient group; understand the research content and sign the informed consent; no family history of mental disorders.

SUMMARY:
This study aims to build a multi-modal collection template and establish a multi-modal database of seven mental disorders including depressive disorders, bipolar disorders, schizophrenia, obsessive-compulsive disorder, anxiety disorders, addictive disorders and sleep-wake disorders by collecting voice information, facial micro-expression, eye tracking, EEG physiology data respectively. This study will contribute to the multi-modal diagnosis of major mental disorders such as depression in the future and realize clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of ICD-11 or DSM-5 for depressive disorders, bipolar disorders, schizophrenia, obsessive-compulsive disorder, anxiety disorders, addictive disorders and sleep-wake disorders, and do not limit subtypes and current disease state;
2. Age 15-60;
3. Han nationality;
4. gender is not limited;
5. have enough audition level to complete the necessary inspection of the research;
6. Understand the research content and sign the informed consent form. If the patient is unable to sign the informed consent form in person due to low education level or other reasons, he or she can be entrusted to sign it by his relatives or his guardian.

Exclusion Criteria:

1. Mental retardation that significantly affects the patient's current mental state;
2. Patients who have serious physical diseases, and it is difficult to complete the necessary examination, including the history of brain trauma or cerebrovascular disease, severe liver cirrhosis, acute and chronic real failure, severe diabetes, aplastic anemia, moderate and severe malnutrition, other serious physical diseases such as nervous system, heart, liver, kidney, endocrine system and blood system, or diseases that may interfere with the test evaluation (abnormal indexes are more than 2 times higher than normal).

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients in Shanghai Mental Health Center; meet ICD-11 or DSM-5 diagnosis of depressive disorders, bipolar disorders, schizophrenia, obsessive-compulsive disorder, anxiety disorders, addictive disorders and sleep-wake disorders (do not limit subtypes and current disease state); age ≥15 years and < 60 years; gender is not limited.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Building a multi-modal database of major mental disorders | at August 2025
  Establish a prediction model by using machine learning methods and build a multi-modal database of major mental disorders to realize the multi-modal diagnosis and curative effect prediction markers for guiding accurate treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, Doctorate, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The project team provides a multimodal data acquisition platform, establishes a shared data management committee, formulates data sharing mechanisms, and defines the rights and obligations of data contributors, data beneficiaries, and the multimodal information system.

REFERENCES:
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Huang Y, Wang Y, Wang H, Liu Z, Yu X, Yan J, Yu Y, Kou C, Xu X, Lu J, Wang Z, He S, Xu Y, He Y, Li T, Guo W, Tian H, Xu G, Xu X, Ma Y, Wang L, Wang L, Yan Y, Wang B, Xiao S, Zhou L, Li L, Tan L, Zhang T, Ma C, Li Q, Ding H, Geng H, Jia F, Shi J, Wang S, Zhang N, Du X, Du X, Wu Y. Prevalence of mental disorders in China: a cross-sectional epidemiological study. Lancet Psychiatry. 2019 Mar;6(3):211-224. doi: 10.1016/S2215-0366(18)30511-X. Epub 2019 Feb 18. PMID 30792114
- [Background] Phillips MR, Zhang J, Shi Q, Song Z, Ding Z, Pang S, Li X, Zhang Y, Wang Z. Prevalence, treatment, and associated disability of mental disorders in four provinces in China during 2001-05: an epidemiological survey. Lancet. 2009 Jun 13;373(9680):2041-53. doi: 10.1016/S0140-6736(09)60660-7. PMID 19524780
- [Background] Kessler RC, Avenevoli S, Costello J, Green JG, Gruber MJ, McLaughlin KA, Petukhova M, Sampson NA, Zaslavsky AM, Merikangas KR. Severity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication Adolescent Supplement. Arch Gen Psychiatry. 2012 Apr;69(4):381-9. doi: 10.1001/archgenpsychiatry.2011.1603. PMID 22474106
- [Background] Rominger A, Cumming P, Brendel M, Xiong G, Zach C, Karch S, Tatsch K, Bartenstein P, la Fougere C, Koch W, Pogarell O. Altered serotonin and dopamine transporter availabilities in brain of depressed patients upon treatment with escitalopram: A [123 I]beta-CIT SPECT study. Eur Neuropsychopharmacol. 2015 Jun;25(6):873-81. doi: 10.1016/j.euroneuro.2014.12.010. Epub 2015 Jan 5. PMID 25819144
- [Background] Gunaratne P, Lloyd AR, Vollmer-Conna U. Mood disturbance after infection. Aust N Z J Psychiatry. 2013 Dec;47(12):1152-64. doi: 10.1177/0004867413503718. Epub 2013 Sep 20. PMID 24056922
- [Background] Merikangas KR, Swendsen J, Hickie IB, Cui L, Shou H, Merikangas AK, Zhang J, Lamers F, Crainiceanu C, Volkow ND, Zipunnikov V. Real-time Mobile Monitoring of the Dynamic Associations Among Motor Activity, Energy, Mood, and Sleep in Adults With Bipolar Disorder. JAMA Psychiatry. 2019 Feb 1;76(2):190-198. doi: 10.1001/jamapsychiatry.2018.3546. PMID 30540352
- [Background] Haque A, Milstein A, Fei-Fei L. Illuminating the dark spaces of healthcare with ambient intelligence. Nature. 2020 Sep;585(7824):193-202. doi: 10.1038/s41586-020-2669-y. Epub 2020 Sep 9. PMID 32908264